CLINICAL TRIAL: NCT05760963
Title: Which Approach to Favor for Ultrasound-guided Lumbar Plexus Block (BPLE). Comparative Study.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN782021/CHUSTE
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2021-04

CONDITIONS: Volunteers
Keywords: Lumbar plexus; ultrasound guided; Trident; Shamrock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult with lumbar echography indication: Adult with lumbar echography indication will be included.
  Interventions: Other: Collection of datas

INTERVENTIONS:
Other: Collection of datas — Analysis lumbar echographies results by Trident ans Shamrock techniques.
  Costiform processes on T12 to L5 were spotted and noted. For Trident technique, quality of image, depth of lumbar plexus and presence of vessels were noted.
  Shamrock technique was performed, the projection of C line (line obtained with a probe put on the iliac crest) was noted with the invisible ink pen. Then the probe was oriented cephalically (for line >C) and caudally (line <C). For each lines, quality of image, depth of lumbar plexus and presence of vessels were also noted.
  The projections of C, >C, <C on the costiform processes were noted.

SUMMARY:
Lumbar plexus block is described as a difficult block, thus requiring experienced practitioners. Many techniques have been used to date, notably anatomical landmarks, neurostimulation, and ultrasound-guided techniques. Among ultrasound-guided techniques, the "Trident" technique was described in 2006, while the "Shamrock" technique was described in 2013. Trident consists in putting the probe sagittally next to the lumbar spine and injecting local anesthetic around the lumbar plexus inside the psoas muscle at the level of L4. It is an out-of-plane puncture.

Shamrock puts the probe transversely on the iliac crest. Authors of the 2013 article said the image obtained with this technique was an image of L4. This technique allows an in-plane puncture, which is a safe technique.

DETAILED DESCRIPTION:
This study aims at describing the level obtained with Shamrock, as well as at comparing depth of lumbar plexus, image quality and presence of vessels between the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult with indication of lumbar echography

Exclusion Criteria:

* Antecedent of spine surgery or spinal malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with indication of lumbar echography will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Projection of line C on the costiform processes | Day: 0
  Analysis by trident techniques results.

SECONDARY OUTCOMES:
Depth of lumbar plexus | Day: 0
  Analysis by trident and shamrock techniques results.
image quality | Day: 0
  Analysis by trident and shamrock techniques results.
presence of vessels | Day: 0
  Analysis by trident and shamrock techniques results.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime WODEY, resident, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No